CLINICAL TRIAL: NCT02514148
Title: Biobehavioral Physical Therapy Strategies Based on Therapeutic Exercise Applied to Chronic Migraine Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Madrid (Other)
Responsible Party: Principal Investigator, Paula Kindelan, Associate Professor, Universidad autónoma de Madrid, Universidad Autonoma de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSEULS-PI-002/2013
Record Dates: First submitted 2015-05-14; First posted 2015-08-03 (Estimated); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Chronic Migraine; Chronic Headache
Keywords: patient education; therapeutic exercise; manual therapy
MeSH Terms: conditions — Headache Disorders | interventions — Exercise Therapy; Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- NO Intervention Control group (Other): No therapeutic intervention are being giving to the group of patients, they only will have their Neurologist previously prescribed pharmacological treatment.
  Interventions: Other: No intervention
- Therapeutic exercise( TE) (Experimental): The intervention giving to the patients consist on a therapeutic exercise protocol based on neck and low intensity general exercises.
  Interventions: Other: Therapeutic exercise
- Therapeutic patient education ( TPE) (Experimental): The intervention giving to the patients consist on a therapeutic patient education based on pain neurophysiology protocol.
  Interventions: Behavioral: Therapeutic patient education
- TE + TPE (Experimental): The intervention giving to the patients consist on the combination of the therapeutic exercise protocol and the therapeutic patient education protocol.
  Interventions: Behavioral: Therapeutic patient education; Other: Therapeutic exercise
- TE + TPE + Manual therapy (Experimental): The intervention giving to the patients consist on the combination of the therapeutic exercise protocol and the therapeutic patient education protocol plus a manual therapy techniques protocol.
  Interventions: Behavioral: Therapeutic patient education; Other: Therapeutic exercise; Other: Manual Therapy

INTERVENTIONS:
Behavioral: Therapeutic patient education — Therapeutic patient education based on pain physiology from a biobehavioral perspective adding a training in coping strategies.
  Other Names: TPE
  Arms: TE + TPE; TE + TPE + Manual therapy; Therapeutic patient education ( TPE)
Other: Therapeutic exercise — Therapeutic exercise consist on stretch of cervical-scapular muscles ( Trapezius and angular of the scapula), Cranium-cervical flexor stabilization exercise, auto cervical tractions, shoulders rotation, low intensity exercise ( walking), craniocervical extension, cervical flexion and extension.
  Other Names: TE
  Arms: TE + TPE; TE + TPE + Manual therapy; Therapeutic exercise( TE)
Other: No intervention — No intervention consist on measure the whole variables in chronic migraine patients to compare it with experimental interventions
  Other Names: NI
  Arms: NO Intervention Control group
Other: Manual Therapy — Manual therapy consist on ; oscillatory traction , maintained craniocervical traction, upper cervical flexion mobilization, side glide roll, anterior-posterior upper cervical mobilization with wedge, lateral glide at the C1-C2 and C2-C3 levels, retraction technique, trigeminocervical neural mobilization , and upper cervical traction, followed by posterior-anterior glide at C4.
  Other Names: MT
  Arms: TE + TPE + Manual therapy

SUMMARY:
The purpose of this study is to know wich combination of treatments are the most effective in patients with chronic migraine. The study design is a simple blind randomized controlled trial (outcomes assessor). The study population: Men and women aged from 18 to 70 years old with chronic migraine for at least 12 weeks. Interventions: A combination of techniques during 6 weeks (6 sessions; 1 per week)

DETAILED DESCRIPTION:
Migraine is a neurological disease characterized by attacks of pulsating headache on one side of the head, presenting autonomic nervous system disfunction. Migraine is associated to significant personal and social burden. Physical activity could worsen patient´s symptoms. Migraine is associated with nausea, vomiting, photophobia and phonophobia Chronic migraine patients according to the third IHS ( International Headache Society) classification suffer headache at least 15 days per month no less than 3 months.

According to Pozo-Rosich et al., migraine incidence worldwide is 2% of the general population. In the US the 18% of migraine patients are females corresponding the 6% to males.

As comorbid diseases usually associated to migraine are found disability, depression, anxiety and biobehavioral disorders. Migraine is a chronic disease which cause biopsychosocial damage and decrease quality of life in its patients. Risk factors to endure Migraine are sex (females), obesity and overuse of headache medicaments.

Migraine origin and its physiopathology in unknown although there are several studies that support a central sensitization mechanism at the level of trigeminocervical complex to explain migraine. Trigeminocervical complex is made by the convergence between superior neurons of the trigeminal nucleus caudalis and the dorsal cervical horns of the first and second cervical levels.

Some authors suggest that it is a biobehavioral disorder that results from a cortical hypersensitivity and an associated social learning process. Behavioral habits and medication intake due to migraine attacks are important factors to keep in mind. Stanos et al. concluded that the best treatment for chronic migraine was a multidisciplinary treatment including biobehavioral and pharmacological approaches. Biobehavioral treatments (BBTs) for chronic pain patients includes therapeutic patient education (TPE) and selfcare, cognitive behavioral interventions, and biobehavioral training (biofeedback, relaxation training, and stress management).

TPE provides contact between the care providers and patients. TPE has been extensively studied in the management of anxiety, stress, and pain for chronic lower back pain. It is thought that in chronic diseases, TPE should be adapted to the needs of patients and caregivers. BBTs were identified as "grade A" evidence in the American Consortium of Evidence Based Headache Guidelines. It has been proposed that BBT based on educational approaches be used to manage migraines.

ELIGIBILITY:
Inclusion Criteria:

* subjects diagnosed with chronic migraine
* Neck, shoulder or spine pain for at least 12 weeks
* Continuous headache may be chronic daily headache or tension headache
* Patients having the willing to undergo the treatment

Exclusion Criteria:

* Patients undergoing physical another therapy treatment in cervical or head areas.
* Patient with degenerative neurological syndrome or fibromyalgia
* Patients with severe cognitive impairment
* Patients undergo any neck, head or shoulder surgical process

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2015-09; Primary Completion 2018-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Quality of Life measured by the HIT-6 Questionnaire | Baseline
  A generic concept reflecting concern with the modification and enhancement of life attributes, e.g., physical, political, moral and social environment; the overall condition of a human life.

SECONDARY OUTCOMES:
Cervical range of Motion measured by CROM ( cervical range of motion device) | Baseline , 6 weeks, 2 months, 4 months, 6 months, one year
  The distance and direction to which a bone joint can be extended. Range of motion is a function of the condition of the joints, muscles, and connective tissues involved. Joint flexibility can be improved through appropriate MUSCLE STRETCHING EXERCISES.
Temporal Summation measured by Von Frey filament | Baseline , 6 weeks, 2 months, 4 months, 6 months, one year
  Postsynaptic Potential Summation: Physiological integration of multiple SYNAPTIC POTENTIAL signals to reach the threshold and initiate postsynaptic ACTION POTENTIALS. In spatial summation stimulations from additional synaptic junctions are recruited to generate s response. In temporal summation succeeding stimuli signals are summed up to reach the threshold. The postsynaptic potentials can be either excitatory or inhibitory (EPSP or IPSP).)
Sleep Disorders measured by Latineen index score | Baseline , 6 weeks, 2 months, 4 months, 6 months, one year
  Conditions characterized by disturbances of usual sleep patterns or behaviors. Sleep disorders may be divided into three major categories: DYSSOMNIAS (i.e. disorders characterized by insomnia or hypersomnia), PARASOMNIAS (abnormal sleep behaviors), and sleep disorders secondary to medical or psychiatric disorders
Medication Adherence scored by a medication calendar | Baseline , 6 weeks, 2 months, 4 months, 6 months, one year
  Voluntary cooperation of the patient in taking drugs or medicine as prescribed. This includes timing, dosage, and frequency
Cope (Adaptation, Psychological) measured by CADC questionnaire ( Adaptation of the Chronic Pain self-efficacy Scale) and CAD- R questionnaire | Baseline , 6 weeks, 2 months, 4 months, 6 months, one year
  A state of harmony between internal needs and external demands and the processes used in achieving this condition
Anxiety measured by EUROQOL score | Baseline , 6 weeks, 2 months, 4 months, 6 months, one year
  Feeling or emotion of dread, apprehension, and impending disaster but not disabling as with ANXIETY DISORDERS.
Catastrophization measured by PCS ( Pain Catastrophizing Scale) | Baseline , 6 weeks, 2 months, 4 months, 6 months, one year
  Cognitive and emotional processes encompassing magnification of pain-related stimuli, feelings of helplessness, and a generally pessimistic orientation.
Phobic Disorders measured by Chronic Pain self-efficacy Scale, BECK | Baseline , 6 weeks, 2 months, 4 months, 6 months, one year
  Anxiety disorders in which the essential feature is persistent and irrational fear of a specific object, activity, or situation that the individual feels compelled to avoid. The individual recognizes the fear as excessive or unreasonable.
Disability Evaluation measured by neck disability Index and CF-PDI ( Craniofacial pain and disability inventory) | Baseline , 6 weeks, 2 months, 4 months, 6 months, one year
  Determination of the degree of a physical, mental, or emotional handicap. The diagnosis is applied to legal qualification for benefits and income under disability insurance and to eligibility for Social Security and workmen's compensation benefits.
  Determination of the degree of a physical, mental, or emotional handicap. The diagnosis is applied to legal qualification for benefits and income under disability insurance and to eligibility for Social Security and workmen's compensation benefits.
  Determination of the degree of a physical, mental, or emotional handicap. The diagnosis is applied to legal qualification for benefits and income under disability insurance and to eligibility for Social Security and workmen's compensation benefits.
Self Efficacy measured by Chronic Pain self-efficacy Scale | Baseline , 6 weeks, 2 months, 4 months, 6 months, one year
  Cognitive mechanism based on expectations or beliefs about one's ability to perform actions necessary to produce a given effect. It is also a theoretical component of behavior change in various therapeutic treatments.
Pain perception outcome assessed by VAS | Baseline , 6 weeks, 2 months, 4 months, 6 months, one year
  The process by which PAIN is recognized and interpreted by the brain.
Quality of Life measured by the HIT-6 Questionnaire | Baseline , 6 weeks, 2 months, 4 months, 6 months, one year
  A generic concept reflecting concern with the modification and enhancement of life attributes, e.g., physical, political, moral and social environment; the overall condition of a human life.
Physical activity measured by IPAQ ( International physical Activity questionnaire) | Baseline , 6 weeks, 2 months, 4 months, 6 months, one year
  The performance of the basic activities of self care or sport such as dressing, ambulation, eating, walking or practicing sports.
Pain Threshold measured by algometer | Baseline , 6 weeks, 2 months, 4 months, 6 months, one year
  Amount of stimulation required before the sensation of pain is experienced.
Pain behaviour assessed by PBQ questionnaire ( Pain behaviour questionnaire) | Baseline , 6 weeks, 2 months, 4 months, 6 months, one year
  The process by which PAIN is recognized and interpreted by the brain.
Kinesiophobia measured by TSK ( Tampa Scale of Kinesiophobia) | Baseline , 6 weeks, 2 months, 4 months, 6 months, one year
  Fear of having a painfull experience due to mevement

CONTACTS AND LOCATIONS:
Overall Officials: Paula Kindelan, MSc, Principal Investigator — associate professor Universidad Autónoma de Madrid
Locations (1):
- Unidad de Ciencias Neurológicas, Madrid, Spain

REFERENCES:
- [Background] Latimer KM. Chronic headache: stop the pain before it starts. J Fam Pract. 2013 Mar;62(3):126-33. PMID 23520582
- [Background] Pozo-Rosich P. [Chronic migraine: its epidemiology and impact]. Rev Neurol. 2012 Apr 10;54 Suppl 2:S3-11. Spanish. PMID 22532240
- [Background] Bashir A, Lipton RB, Ashina S, Ashina M. Migraine and structural changes in the brain: a systematic review and meta-analysis. Neurology. 2013 Oct 1;81(14):1260-8. doi: 10.1212/WNL.0b013e3182a6cb32. Epub 2013 Aug 28. PMID 23986301
- [Background] Volcy M, Sheftell FD, Tepper SJ, Rapoport AM, Bigal ME. Tinnitus in migraine: an allodynic symptom secondary to abnormal cortical functioning? Headache. 2005 Sep;45(8):1083-7. doi: 10.1111/j.1526-4610.2005.05193_2.x. PMID 16109127
- [Background] Calhoun AH, Ford S, Millen C, Finkel AG, Truong Y, Nie Y. The prevalence of neck pain in migraine. Headache. 2010 Sep;50(8):1273-7. doi: 10.1111/j.1526-4610.2009.01608.x. Epub 2010 Jan 18. PMID 20100298
- [Background] Headache Classification Committee of the International Headache Society (IHS). The International Classification of Headache Disorders, 3rd edition (beta version). Cephalalgia. 2013 Jul;33(9):629-808. doi: 10.1177/0333102413485658. No abstract available. PMID 23771276
- [Background] Lipton RB, Bigal ME, Diamond M, Freitag F, Reed ML, Stewart WF; AMPP Advisory Group. Migraine prevalence, disease burden, and the need for preventive therapy. Neurology. 2007 Jan 30;68(5):343-9. doi: 10.1212/01.wnl.0000252808.97649.21. PMID 17261680
- [Background] Ruscheweyh R, Muller M, Blum B, Straube A. Correlation of headache frequency and psychosocial impairment in migraine: a cross-sectional study. Headache. 2014 May;54(5):861-71. doi: 10.1111/head.12195. Epub 2013 Aug 23. PMID 23980919
- [Background] Finocchi C, Villani V, Casucci G. Therapeutic strategies in migraine patients with mood and anxiety disorders: clinical evidence. Neurol Sci. 2010 Jun;31 Suppl 1:S95-8. doi: 10.1007/s10072-010-0297-2. PMID 20464594
- [Background] Bartsch T, Goadsby PJ. The trigeminocervical complex and migraine: current concepts and synthesis. Curr Pain Headache Rep. 2003 Oct;7(5):371-6. doi: 10.1007/s11916-003-0036-y. PMID 12946290
- [Background] Grazzi L, Bussone G. What future for treatment of chronic migraine with medication overuse? Neurol Sci. 2011 May;32 Suppl 1:S19-22. doi: 10.1007/s10072-011-0553-0. PMID 21533706
- [Background] Gerber WD, Schoenen J. Biobehavioral correlates in migraine: the role of hypersensitivity and information-processing dysfunction. Cephalalgia. 1998 Feb;18 Suppl 21:5-11. doi: 10.1177/0333102498018s2103. PMID 9533662
- [Background] Stanos S. Focused review of interdisciplinary pain rehabilitation programs for chronic pain management. Curr Pain Headache Rep. 2012 Apr;16(2):147-52. doi: 10.1007/s11916-012-0252-4. PMID 22427179
- [Background] Andrasik F, Buse DC, Grazzi L. Behavioral medicine for migraine and medication overuse headache. Curr Pain Headache Rep. 2009 Jun;13(3):241-8. doi: 10.1007/s11916-009-0041-x. PMID 19457287
- [Background] Carlson CR. Psychological considerations for chronic orofacial pain. Oral Maxillofac Surg Clin North Am. 2008 May;20(2):185-95, vi. doi: 10.1016/j.coms.2007.12.002. PMID 18343324
- [Background] Rains JC, Penzien DB, McCrory DC, Gray RN. Behavioral headache treatment: history, review of the empirical literature, and methodological critique. Headache. 2005 May;45 Suppl 2:S92-109. doi: 10.1111/j.1526-4610.2005.4502003.x. PMID 15921506
- [Background] Daviet JC, Bonan I, Caire JM, Colle F, Damamme L, Froger J, Leblond C, Leger A, Muller F, Simon O, Thiebaut M, Yelnik A. Therapeutic patient education for stroke survivors: Non-pharmacological management. A literature review. Ann Phys Rehabil Med. 2012 Dec;55(9-10):641-56. doi: 10.1016/j.rehab.2012.08.011. Epub 2012 Sep 7. English, French. PMID 23000090
- [Background] Louw A, Diener I, Butler DS, Puentedura EJ. The effect of neuroscience education on pain, disability, anxiety, and stress in chronic musculoskeletal pain. Arch Phys Med Rehabil. 2011 Dec;92(12):2041-56. doi: 10.1016/j.apmr.2011.07.198. PMID 22133255
- [Background] Nicholson R, Nash J, Andrasik F. A self-administered behavioral intervention using tailored messages for migraine. Headache. 2005 Oct;45(9):1124-39. doi: 10.1111/j.1526-4610.2005.00236.x. PMID 16178943
- [Background] Buse DC, Andrasik F. Behavioral medicine for migraine. Neurol Clin. 2009 May;27(2):445-65. doi: 10.1016/j.ncl.2009.01.003. PMID 19289225
- [Background] Kindelan-Calvo P, Gil-Martinez A, Paris-Alemany A, Pardo-Montero J, Munoz-Garcia D, Angulo-Diaz-Parreno S, La Touche R. Effectiveness of therapeutic patient education for adults with migraine. A systematic review and meta-analysis of randomized controlled trials. Pain Med. 2014 Sep;15(9):1619-36. doi: 10.1111/pme.12505. Epub 2014 Aug 26. PMID 25159212